CLINICAL TRIAL: NCT06164249
Title: Quantification of Internal Training Load: Toward the Prediction of the Distribution of Hypertrophy
Brief Title: Quantification of Internal Training Load
Acronym: QUADRATURE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université de Nantes (Other)
Responsible Party: Principal Investigator, Lilian Lacourpaille, Doctor, Université de Nantes
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: EM_LL_2024
Record Dates: First submitted 2023-11-30; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Hypertrophy; Resistance Training; Muscle
Keywords: Muscle activation; Muscle volume; Muscle stress; Muscle mass
MeSH Terms: conditions — Hypertrophy | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Three independent groups :
  * Control (no strengthening)
  * Nordic (strengthening in Nordic Hamstring exercise)
  * Deadlift (strengthening in Deadlift exercise)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator is blind. Participants know in which group they are as each group is composed of no exercise (control), Nordic hamstring exercise (Nordic), or Deadlift exercise (Deadlift)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nordic (Experimental): Training regimens composed of nordic exercise
  Interventions: Other: strength training
- Deadlift (Experimental): Training regimens composed of deadlift exercise
  Interventions: Other: strength training
- Control (No Intervention): Training regimens composed of no exercise

INTERVENTIONS:
Other: strength training — Strength training, three times a week, during nine weeks.
  Arms: Deadlift; Nordic

SUMMARY:
The aim of this study is to determine whether the distribution of internal load predicts the distribution of muscle hypertrophy among hamstring heads after a 10-week resistance exercise program. The hypothesis is that the distribution of internal muscle load among the hamstring is related to the distribution of muscle hypertrophy.

DETAILED DESCRIPTION:
It is well accepted that muscle stress (mechanical and/or metabolic) is the major way to induce muscle hypertrophy. While this link between muscle stress and hypertrophy is pivotal is sport training, prevention and rehabilitation, it remains poorly understood. To date, the only indirect evidence of relationship of muscle stress and muscle hypertrophy is the similar patterns (from independent studies) between muscle damage and hypertrophy within quadriceps (i.e., rectus femoris (RF) > vastus (VL) = vastus medialis VM), hamstring, and triceps surae. However, muscle damage is an indirect proof of muscle mechanical stress. With the quantification of internal muscle load, it is interesting to determine whether the muscle that receives the larger stress exhibits the larger hypertrophy.

ELIGIBILITY:
Inclusion Criteria:

* No history of lower limb injury
* No chronic pathology associated with a long term care

Exclusion Criteria:

* Individual enrolled in a research study

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-01-29 (Estimated); Primary Completion 2024-04-02 (Estimated); Study Completion 2024-05-19 (Estimated)

PRIMARY OUTCOMES:
Muscle volume | 10 weeks
  Hypertrophy
Internal training load | 10 weeks
  Magnitude and onset/offset of muscle activation

SECONDARY OUTCOMES:
Maximal strength Nordic | 10 weeks
  Maximal strength during the Nordic exercise
Maximal strength Deadlift | 10 weeks
  Maximal strength during the Deadlift exercise

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available from a Dryad Digital Repository